CLINICAL TRIAL: NCT04624152
Title: The Combined Effects of Hypoxia and Subconcussive Head Impacts on Neurocognitive Function: a Pilot Randomized Crossover Study
Brief Title: The Role of Hypoxia on Subconcussive Head Impacts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Keisuke Kawata, Assistant Professor Kinesiology, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1806106387
Record Dates: First submitted 2020-11-02; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Trauma, Brain
Keywords: soccer heading; subconcussive head impacts; hypoxia
MeSH Terms: conditions — Brain Injuries, Traumatic; Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normobaric Hypoxia (Experimental): Large weather balloons will be filled with a normobaric hypoxic inspirate (FiO2 = 0.15) produced by a nitrogen generator (CAT 12; Colorado Altitude Training, Boulder, CO) to simulate an altitude of 2600 m (8500 ft). Participants breathed this inspirate through a two-way non-rebreathing valve (2700; Hans Rudolph, Kansas City, KS) and an oronasal mask (7450 V2; Hans Rudolph, Kansas City, KS).
  Participants breathed this inspirate from 15 minutes before the pre-heading time point until the conclusion of the 0h post-heading time point.
  Interventions: Behavioral: Soccer heading
- Normobaric Normoxia (Placebo Comparator): Large weather balloons will be filled with room air (FiO2 = 0.21). Participants breathed this normobaric normoxic inspirate through a two-way non-rebreathing valve (2700; Hans Rudolph, Kansas City, KS) and an oronasal mask (7450 V2; Hans Rudolph, Kansas City, KS).
  Participants breathed this inspirate from 15 minutes before the pre-heading time point until the conclusion of the 0h post-heading time point.
  Interventions: Behavioral: Soccer heading

INTERVENTIONS:
Behavioral: Soccer heading — A standardized and reliable soccer heading protocol will be used to induce subconcussive impacts for the experiment. A triaxial accelerometer (Triax Technologies, Norwalk, CT) embedded in a head-band pocket and positioned back of the head to monitor linear and rotational head accelerations. A JUGS soccer machine (JUGS Sports, Tualatin, OR) will be used to simulate a soccer throw-in with a standardized ball speed of 25 mph across all groups. The ball speed is similar to when soccer players make a long throw-in from the sideline to mid-field. Soccer players frequently perform this maneuver during practices and games. Participants will stand approximately 40ft away from the machine to perform the heading. Participants will perform a total of 10 headers at a rate of 1 header per minute and will be instructed to direct the ball back towards the JUGS machine. Previous uses of this soccer heading model have reported an average peak linear acceleration per header of 14.5 to 33.5 g.

SUMMARY:
The purpose of this study is to examine the combined effects of hypoxia and a short bout of subconcussive head impacts on neurocognitive and ocular-motor function and plasma expression of brain-derived blood biomarkers.

DETAILED DESCRIPTION:
The purpose of the pilot study is to observe preliminary trends in neural response to subconcussive head impacts in hypoxic condition. This work will provide a critical un-tested knowledge regarding the combined effects of subconcussion and hypoxic condition (mimicking high altitude), which will be used in our upcoming grant proposal to the Department of Defense (DoD). Military personnel, particularly those who are deployed to Afghanistan, are constantly subjected to hypoxic condition, given that the majority of military land operations in Afghanistan occur at 2000-3000 meters (6500-10,000 feet). This level of altitude does not elicit major side effects, yet neural functions may experience some degree of perturbation (i.e., slowed reaction time, altered night vision). Concurrently, these military personnel, who operate at high altitudes, often incur subconcussive forces to the head. These subconcussive head impacts can be induced by exposure to, for example, flash-bang grenades, artillery fire, recoilless rifle, improvised explosive devices (IEDs), and head collision. The combined effects of these two stressors have the potential to attenuate one's readiness, operational efficiency, and overall brain function, but the combined effects have never been studied to date. As a result, one of four study topics that the Defense Centers of Excellence deems urgent is: Document the effects of altitude exposure on mild traumatic brain injury (mTBI) and blast-induced neurotrauma (BINT). To answer the question, we hypothesized that there will be an exponential worsening in neurocognitive function and in ocular-motor system functioning, and increased plasma expression of brain-derived biomarkers, after subconcussive head impacts under hypoxic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 26 years old
* Current or former soccer player (i.e., collegiate, intramural, club, professional)
* At least 3 years of soccer heading experience
* Participants can read and speak English
* Participants have cell phone or computer with internet access to schedule for follow-up visits via email or text message
* Participant is willing to refrain from participating in any sport activity that purposefully uses one's head to maneuver (American football, ice-hockey, rugby, wrestling, and soccer heading) during study participation

Exclusion Criteria:

* Any head, neck, or face injury in the 1 year prior to the study (e.g., concussion, eye injury)
* History of vestibular, ocular, or vision dysfunction (e.g., macular degeneration)
* Currently taking any medications that trigger drowsiness
* Pregnancy
* Any history of neurological disorders (e.g., seizure disorders, closed head injuries with loss of consciousness greater than 15 minutes, CNS neoplasm, spinal cord injury/surgery, history of stroke)
* Lower extremity injury that would prohibit normal walking
* Metal implants in the head

Conditional Exclusion Criteria

Based on participants' self report: those who meet any of the following criteria, he/she will be either excluded or rescheduled (if they still wish to participate in the study):

* Slept less than 4 hours during the night prior to the testing day
* Consumed more than 3 alcoholic drinks within 24h prior to testing
* Used recreational drugs 24h prior to the testing day
* Consumed more than 300 mg of caffeine (the equivalent of about 3 cups of coffee) within 1h before testing sessions

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — As a part of the neurocognitive assessment, participants self-select one of the gender options from a list.
Enrollment: 10 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Acute change in neurocognitive function from pre-heading at 0 hour post-heading | Neurocognitive function will be assessed at pre- and 0 hour post-heading
  Participants will complete a computerized neurocognitive assessment (Immediate Post-Concussion Assessment and Cognitive Testing).
Acute change in convergence function from pre-heading at 0 hour post-heading | Conversion function will be assessed at pre- and 0 hour post-heading
  Participants will undergo near-point of convergence (in centimeter) to evaluate how closely one can visualize a moving target without double vision occurs.
Acute change in brain-derived blood biomarkers from pre-heading at 0 hour post-heading | Blood samples will be collected at pre- and 0 hour post-heading
  Blood samples will be collected and centrifuged at 1500 x g for ten minutes at 4 degree celsius. Plasma will be aliquoted and stored at -80 degree celsius until analysis.
  Plasma samples will be assayed for neurofilament-light (NfL), glial fibrillary acidic protein (GFAP), and tau.

SECONDARY OUTCOMES:
Change in neurocognitive function at 24 hours post-heading follow-up | Neurocognitive function will also assessed at 24 hours post-heading
  Upon their return to the laboratory, participants will again complete a computerized neurocognitive assessment (Immediate Post-Concussion Assessment and Cognitive Testing).
Change in ocular-motor function at 24 hours post-heading follow-up | Ocular-motor function will also assessed at 24 hours post-heading
  Upon their return to the laboratory, participants will again undergo three ocular-motor assessments: 1) near-point of convergence; 2) King-Devick Test--a brief assessment of saccadic eye movements, attention, and visual and language processing; and 3) the EYE-SYNC smooth pursuit task.
Change in brain-derived blood biomarkers at 24 hours post-heading follow-up | A third blood sample will be collected at 24 hours post-heading
  Blood samples will be collected and centrifuged at 1500 x g for ten minutes at 4 degree celsius. Plasma will be aliquoted and stored at -80 degree celsius until analysis.
  Plasma samples will be assayed for neurofilament-light (NfL), glial fibrillary acidic protein (GFAP), and tau.
Acute change in saccadic eye movement function from pre-heading at 0 and 24 hour post-heading | Saccadic eye movement function will be assessed at pre- , 0, and 24 hour post-heading
  Participants will undergo King-Devick Test--a brief assessment of saccadic eye movements, attention, and visual and language processing
Acute change in smooth eye pursuit function from pre-heading at 0 and 24 hour post-heading | Smooth eye pursuit function will be assessed at pre- , 0, and 24 hour post-heading
  Participants will undergo the EYE-SYNC smooth pursuit task.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Bloomington, Indiana, United States